CLINICAL TRIAL: NCT03579641
Title: Precision Event Monitoring for Patients With Heart Failure Using HeartLogic: PREEMPT-HF
Brief Title: Precision Event Monitoring for Patients With Heart Failure Using HeartLogic
Acronym: PREEMPT-HF
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PREEMPT-HF
Record Dates: First submitted 2018-06-04; First posted 2018-07-06 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Defibrillators, Implantable; Monitoring, Physiologic; Cardiac Resynchronization Therapy; Cardiovascular Disease; Heart Disease
Keywords: Heart Failure; Implantable Cardioverter Defibrillator; Cardiac Resynchronization Therapy Defibrillator; Heart Failure Sensor Data; 30-day Heart Failure Readmission; Ventricular Tachycardia/Ventricular Fibrillation Therapy; Non-Heart Failure Hospitalization; HeartLogic Feature; Latitude Remote Patient Monitor; Data Linkage; Sleep Incline Sensor; Respiratory Sensor; Decongestive Intravenous therapy; Decompensation
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Heart Diseases; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Implantable Cardiac device with HeartLogic feature: Patients with Heart Failure, implanted with Boston Scientific Implantable Cardioverter Defibrillator or Defibrillator with Cardiac Resynchronization device with HeartLogic feature
  Interventions: Device: HeartLogic Sensors

INTERVENTIONS:
Device: HeartLogic Sensors — HeartLogic Sensors

SUMMARY:
The goal of the PREEMPT-HF study is to collect device and clinical event data to evaluate extended applications of the HeartLogic Heart Failure Diagnostic (HeartLogic) in a broad spectrum of heart failure patients with an implantable cardioverter defibrillator or cardiac resynchronization therapy defibrillator. There are no primary safety and/or efficacy endpoints for this study.

Heart failure is a complex clinical syndrome with high morbidity, mortality, and economic burden. Chronic Heart Failure is persistent, gradually progressive, and punctuated by episodes of acute worsening leading to hospitalizations. Therefore, there remains an unmet clinical need to slow the progression of Heart Failure and prevent hospitalizations. HeartLogic, available in Boston Scientific cardiac resynchronization therapy devices and defibrillators, combines novel sensor parameters such as heart sounds and respiration with other measurements like thoracic impedance, heart rate, and activity into a HeartLogic Index for the early detection of worsening Heart Failure. However, there is limited data on the association of HeartLogic with the risk of Hear Failure readmissions and tachyarrhythmias, or for phenotyping the broad spectrum of Heart Failure patients.

DETAILED DESCRIPTION:
Subjects will be followed for approximately 12 months after the baseline visit to collect the required number of clinical events to support the study objectives. These events are called Reviewable Clinical Events, and include all-cause hospitalizations and Heart Failure outpatient visits.

Clinical event definitions are as follows:

* Hospitalization (all-cause): the subject is admitted to inpatient hospital care and discharged on a different calendar date.
* Heart Failure Hospitalization: the subject is admitted with signs/symptoms of congestive heart failure and receives unscheduled augmented Heart Failure therapy with oral or intravenous medications, ultrafiltration therapy or other parenteral therapy.
* Heart Failure Readmission (30-day): the subject is admitted for an unplanned hospitalization for any cause within 30 days post discharge from a Heart Failure hospitalization.
* Heart Failure Outpatient Visit: the subject has signs/symptoms of Congestive Heart Failure, and receives unscheduled intravenous decongestive therapy (e.g., Intravenous diuretics, Intravenous inotropes, Intravenous vasoactive drugs, ultrafiltration) in a setting that does not involve a hospitalization (e.g., emergency room, Heart Failure clinic, primary care clinic, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 or above, or of legal age to give informed consent specific to each country and national laws.
* Subject has a documented diagnosis of heart failure.
* Subject has a Boston Scientific Cardiac Resynchronization Therapy Defibrillator or Implantable Cardioverter Defibrillator device implant that has HeartLogic, with Heart Failure Sensors turned ON, Respiratory Sensor turned ON, and Sleep Incline Sensor turned ON.
* Subject has an active bipolar right ventricle lead implant.
* Subject is enrolled in LATITUDE (NXT 5.0 or future version), and is willing to be remotely monitored from the baseline visit for approximately 12 months with HeartLogic disabled.

Exclusion Criteria:

* Subject has received or is scheduled to receive a heart transplant or ventricular assist device (VAD).
* Subject is enrolled in any concurrent clinical study without prior Boston Scientific written approval (excluding registries).
* Subject has a life expectancy of less than 12 months.
* Subject has a history of non-compliance to medical care or known inability to comply with requirements of the clinical study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Heart Failure implanted with Boston Scientific Cardiac Resynchronization Therapy Defibrillator or Implantable Cardioverter Defibrillator using HeartLogic
Sampling Method: Non-Probability Sample
Enrollment: 2184 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Association of HeartLogic sensors with 30-day HF re-admission | Heartlogic sensor data will be evaluated for the association to HF re-admission during the 30 days after the index event (e.g. the first HF hospitalization that occurs during the trial).
  To compare a mean sensor value change (admission - discharge) between the no-readmission group and the 30-day readmission group.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gaertner, Study Director — Boston Scientific Corporation
Locations (88):
- United States (56):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cardiology Associates of Northeast Arkansas, Jonesboro, Arkansas
  - Baptist Health Medical Center (Little Rock), Little Rock, Arkansas
  - Providence St. Joseph Medical Center, Burbank, California
  - Mission Hospital, Mission Viejo, California
  - Stanford University Medical Center, Stanford, California
  - Harbor UCLA Medical Center, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Cardiology Physicians, PA, Newark, Delaware
  - Baptist Medical Center, Jacksonville, Florida
  - Watson Clinic Center for Research, Inc., Lakeland, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Florida Hospital, Winter Park, Florida
  - CorVita Science Foundation (NFP), Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland Medical System, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Mass Heart and Rhythm, Leominster, Massachusetts
  - Advanced Cardiovascular Clinic, Flint, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Luke's Hospital-Duluth, Duluth, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - Heart and Vascular Hattiesburg Clinic, Hattiesburg, Mississippi
  - St. Joseph Mercy Hospital Oakland, Pontiac, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Capital Cardiology Associates, Albany, New York
  - Columbia University Medical Center, New York, New York
  - Strong Memorial Hospital of the University of Rochester, Rochester, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Southern Oregon Cardiology, LLC, Medford, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - St. Francis Health System - St. Francis Hospital, Greenville, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seton Medical Center, Austin, Texas
  - The University of Texas, Southwestern Medical Center, Dallas, Texas
  - Orion Medical, Pasadena, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Riverside Regional Medical Center, Newport News, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
- Prince Charles Hospital, Chermside, Australia
- OLVZ Aalst, Aalst, Belgium
- Canada (2):
  - CHUM, Montreal
  - IUCPQ, Ste-Foy
- Aarhus University Hospital, Aarhus, Denmark
- France (4):
  - CHU de Caen, Caen
  - CHU de Nantes - Hôpital Laennec, Nantes
  - APHP - Hospital de la Pitie-Salpetriere, Paris
  - CHU de St. Etienne, Saint-Priest-en-Jarez
- Germany (2):
  - Augusta Kranken Anstalt GmbH - Klinik für Kardiologie und Angiologie, Bochum
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
- Hong Kong (3):
  - Grantham Hospital, Aberdeen
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- University Hospital Waterford, Waterford, Ireland
- Italy (4):
  - Az. Osp. G. Ciaccio Pontepiccolo, Catanzaro
  - Az. Osp. Monaldi, Naples
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Azienda Osp Univ Integrata di Verona, Verona
- Netherlands (3):
  - AMC, Amsterdam
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum, Utrecht
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de Gran Canaria Dr. Negrin, Las Palmas
  - Hospital Universitario Virgen De La Victoria, Málaga
- United Kingdom (7):
  - Belfast City Hospital, Belfast
  - Golden Jubilee National Hospital, Clydebank
  - Ninewells Hospital and Medical School, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - South Manchester University Hospital Trust, Manchester
  - Northern General Hospital, Sheffield
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Ambrosy AP, Fonarow GC, Butler J, Chioncel O, Greene SJ, Vaduganathan M, Nodari S, Lam CSP, Sato N, Shah AN, Gheorghiade M. The global health and economic burden of hospitalizations for heart failure: lessons learned from hospitalized heart failure registries. J Am Coll Cardiol. 2014 Apr 1;63(12):1123-1133. doi: 10.1016/j.jacc.2013.11.053. Epub 2014 Feb 5. PMID 24491689
- [Background] Gheorghiade M, Pang PS. Acute heart failure syndromes. J Am Coll Cardiol. 2009 Feb 17;53(7):557-573. doi: 10.1016/j.jacc.2008.10.041. PMID 19215829
- [Background] Boehmer JP, Hariharan R, Devecchi FG, Smith AL, Molon G, Capucci A, An Q, Averina V, Stolen CM, Thakur PH, Thompson JA, Wariar R, Zhang Y, Singh JP. A Multisensor Algorithm Predicts Heart Failure Events in Patients With Implanted Devices: Results From the MultiSENSE Study. JACC Heart Fail. 2017 Mar;5(3):216-225. doi: 10.1016/j.jchf.2016.12.011. PMID 28254128
- [Background] Whellan DJ, Lindenfeld J. Easy to Predict, Difficult to Prevent. JACC Heart Fail. 2017 Mar;5(3):226-228. doi: 10.1016/j.jchf.2017.01.006. No abstract available. PMID 28254129
- [Background] Desai AS. The three-phase terrain of heart failure readmissions. Circ Heart Fail. 2012 Jul 1;5(4):398-400. doi: 10.1161/CIRCHEARTFAILURE.112.968735. No abstract available. PMID 22811548
- [Background] Dharmarajan K, Wang Y, Lin Z, Normand ST, Ross JS, Horwitz LI, Desai NR, Suter LG, Drye EE, Bernheim SM, Krumholz HM. Association of Changing Hospital Readmission Rates With Mortality Rates After Hospital Discharge. JAMA. 2017 Jul 18;318(3):270-278. doi: 10.1001/jama.2017.8444. PMID 28719692
- [Background] Shah SJ, Katz DH, Selvaraj S, Burke MA, Yancy CW, Gheorghiade M, Bonow RO, Huang CC, Deo RC. Phenomapping for novel classification of heart failure with preserved ejection fraction. Circulation. 2015 Jan 20;131(3):269-79. doi: 10.1161/CIRCULATIONAHA.114.010637. Epub 2014 Nov 14. PMID 25398313
- [Derived] Sauer AJ, Stolen CM, Shute JB, Kwan B, Wariar R, Ruble SB, Gardner RS, Boehmer JP. Results of the Precision Event Monitoring for Patients With Heart Failure Using HeartLogic Study (PREEMPT-HF). JACC Heart Fail. 2025 Jun;13(6):973-983. doi: 10.1016/j.jchf.2025.01.028. Epub 2025 Apr 23. PMID 40272337

DOCUMENTS (1):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT03579641/Prot_000.pdf